CLINICAL TRIAL: NCT05989191
Title: An International Field Study for the Reliability and Validity of the EORTC PATSAT-C33 and the EORTC OUT-PATSAT7 Questionnaires
Brief Title: Study for the Reliability and Validity of the EORTC PATSAT-C33 and the EORTC OUT-PATSAT7 Questionnaires
Acronym: PATSAT
Status: Active, not recruiting | Type: Observational
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Other Study IDs: IC 2019-07
Record Dates: First submitted 2020-02-11; First posted 2023-08-14 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Cancer
Keywords: Quality of life; Cancer care pathway; Patient satisfaction; Care improvement
MeSH Terms: conditions — Neoplasms; Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to validate the EORTC PATSAT-C33 and EORTC OUT-PATSAT7 questionnaires scale structure in a large international field study.

DETAILED DESCRIPTION:
Patient satisfaction is now recognized as an important indicator of care quality. Measures of patient satisfaction with care can facilitate monitoring initiatives for care improvement over time. The EORTC Quality of Life Group has cross-culturally validated a stand-alone in-patient satisfaction with cancer care questionnaire, the IN-PATSAT32. Advances in cancer care delivery required further development of this questionnaire to assess patients' perceived quality of the care received in outpatient cancer care settings. Phase I to III of this process have been completed, resulting in the EORTC PATSAT-C33 satisfaction with cancer care core questionnaire to assess cancer care delivery as a whole and the complementary EORTC OUT-PATSAT7, a questionnaire for the specific outpatient care settings. These questionnaires concern all patients treated for their cancer, in the assessed service, regardless of the stage and type of cancer.

ELIGIBILITY:
Inclusion Criteria:

Patients regardless of cancer site or stage of disease (i.e. local, loco-regional, metastatic, in remission) will be invited to participate if they meet the following criteria:

1. Diagnosis of cancer confirmed histologically.
2. Patients are 18 years or older (to be adapted for compliance with each country regulation).
3. Patients are willing to express their non-opposition to participate in the study.
4. Patients are able to read and understand the language of questionnaires.
5. Patients have the cognitive ability to complete the questionnaires.
6. Patients have had a sufficient experience of the cancer treatment setting :

   a. For outpatients consulting in a chemotherapy day clinic/consultation for oral treatment, ambulatory radiotherapy or consultation for follow-up surveillance to check for signs of recurrence : i) between 3 to 6 cycles of chemotherapy or at least 2 cycles of other cancer treatment (e.g., biological oral therapy) or ii) between 2 to 6 weeks of radiotherapy or iii) within the 3rd to 24th month post-cancer treatment. b. For inpatients consulting on an oncology or a surgery ward at least 3 days of hospital stay

Exclusion Criteria:

Patients will be excluded if they are :

1. Participating in another patient-reported outcome investigation that may interfere with this study.
2. Experiencing any psychiatric condition or major cognitive impairment that may hamper completion of self-reported questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with cancer care setting as outpatient, chemotherapy day clinic/consultation for oral treatment, ambulatory radiotherapy or consultation for follow-up surveillance or inpatients or surgery ward.
Sampling Method: Non-Probability Sample
Enrollment: 690 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Validate the EORTC PATSAT-C33 questionnaire | At inclusion
  Adequacy of confirmatory factor analyses estimates of EORTC PATSAT-C33 and EORTC OUT-PATSAT7 questionnaires
  PATSAT-C33 scales:
  * D/Technical Skills
  * D/Information Exchange D/Affective Behaviour
  * N/RT Information
  * N/RT Affective Behaviour
  * Coordination
  * Interaction/HCP
  PATSAT-C33 single items :
  * Family involvement
  * Access/parking
  * Access/way
  * Environment
  * Overall care
Validate the EORTC OUT-PATSAT7 questionnaire | At inclusion
  Adequacy of confirmatory factor analyses estimates of EORTC PATSAT-C33 and EORTC OUT-PATSAT7 questionnaires
  OUT-PATSAT7 scales:
  * Convenience
  * Transition
  OUT-PATSAT7 single item
  - Continuity

SECONDARY OUTCOMES:
Cross-cultural applicability and acceptability | At inclusion
  Adequacy of estimates of cross-cultural applicability and acceptability
Reliability including test-retest and internal consistency | change between inclusion and week 2
  Adequacy of estimates for Reliability including test-retest and internal consistency
Validity, including construct (known-group comparisons) | At inclusion
  Adequacy of estimates of validity, including construct (known-group comparisons)
Convergent and divergent validity | At inclusion
  Adequacy of estimates of convergent and divergent validity
Responsiveness to change | change between inclusion and year 1
  Adequacy of estimates of responsiveness to change
Cross-cultural invariance of psychometric properties | At inclusion
  Adequacy of estimates of cross-cultural invariance of psychometric properties

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut Curie, Paris
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bredart A, Kop JL, Shamieh O, Fox L, Alrjoub W, Conroy T, Turhal NS, Arraras IJ, Bultijnck R, Harle A, Van Hemelrijck M, Pinto E, Roth EJU, Ioannidis G, Costantini A, Chalk T, Young T, Rohde G, Ishiki H, Kikawa Y, Schmidt H, Vassiliou V, Shayler S, Marchal F, Amelie A, Lehmann J; EORTC Quality of Life Group. Phase IV international prospective validation of the EORTC patient satisfaction core questionnaire (EORTC PATSAT-C33) and outpatient module (EORTC OUT-PATSAT7). BMC Cancer. 2025 Nov 26;25(1):1824. doi: 10.1186/s12885-025-15119-3. PMID 41299425